CLINICAL TRIAL: NCT06711965
Title: Interactive Design of Patient-Specific Molds for Tissue Shaping
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0265; NCI-2024-09605 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-11-18; First posted 2024-12-02 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Mastectomy
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoperative Use of 3D Printed Breast Mold (Experimental): Participants will be randomized using a 1:1 ration to 1 of 2 conditions
  Interventions: Procedure: Standard of care reconstruction
- Standard of Care Reconstruction (Experimental): Participants will be randomized using a 1:1 ration to 1 of 2 conditions
  Interventions: Procedure: Surgery, Breast Mold

INTERVENTIONS:
Procedure: Standard of care reconstruction — Participants will receive standard of care reconstruction
  Arms: Intraoperative Use of 3D Printed Breast Mold
Procedure: Surgery, Breast Mold — Participants will undergo surgery. The surgeon may utilize the custom breast mold in shaping the autologous tissue flap for particiapnts.
  Arms: Standard of Care Reconstruction

SUMMARY:
The goal of this study is to develop clinical decision-support algorithms for designing participants-specific breast molds for tissue shaping. Autologous breast reconstruction is an important part of breast cancer rehabilitation for many participants. Our goal is to increase the efficiency of autologous breast reconstruction by helping the surgeon design participants-specific molds for shaping tissue into an acceptable breast form.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the efficiency of autologous reconstruction performed with 3D-printed participants-specific breast molds designed using our clinical decision-support algorithms.

Secondary Objectives:

To assess the total number of times the mold was used by the surgeons in the intervention group.

To compare the intraoperative time for shaping tissue in control versus intervention group.

To collect information on the type of revisions for aesthetic purposes required in control versus intervention group.

To assess the number and type of complications experienced in control versus intervention group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. Patients who are willing and able to provide informed consent
3. Patients who are scheduled to undergo breast reconstruction with free flap (Deep Interior Epigastric Artery Perforator (DIEP) flap or Transverse Rectus Abdominis Myocutaneous (TRAM) flap)

Exclusion Criteria:

1. Patients whose surgical plan includes the use of stacked flaps (DIEP + other free flap, usually from the thigh or buttock)
2. Patients whose surgical plan includes the use of DIEP flap with vascularized lymph node transfer
3. Patients undergoing neoadjuvant radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse eEents (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ashleigh M Francis, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org